CLINICAL TRIAL: NCT00025298
Title: A Feasibility Study Of Primary Chemotherapy Followed By Concomitant Chemoradiation With And Without Amifostine In Patients With Locally Advanced Undifferentiated Nasopharyngeal Cancer (UNPC)
Brief Title: Chemotherapy Plus Radiation Therapy With or Without Amifostine in Treating Patients With Locally Advanced Cancer of the Nasopharynx
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-24981; EORTC-24981
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Head and Neck Cancer; Oral Complications; Radiation Toxicity
Keywords: stage II nasopharyngeal cancer; stage III nasopharyngeal cancer; stage IV nasopharyngeal cancer; oral complications; drug/agent toxicity by tissue/organ; radiation toxicity
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Head and Neck Neoplasms; Radiation Injuries; Nasopharyngeal Neoplasms | interventions — Amifostine; Carboplatin; Cisplatin; Paclitaxel; Radiotherapy

INTERVENTIONS:
Drug: amifostine trihydrate
Drug: carboplatin
Drug: cisplatin
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells. Giving chemoprotective drugs such as amifostine may protect normal cells from the side effects of chemotherapy and radiation therapy.

PURPOSE: Randomized phase II trial to compare the effectiveness of paclitaxel and carboplatin followed by cisplatin plus radiation therapy with or without amifostine in treating patients who have locally advanced cancer of the nasopharynx.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall incidence of grade 3 or 4 mucositis in patients with locally advanced undifferentiated nasopharyngeal cancer treated with paclitaxel and carboplatin followed by cisplatin and radiotherapy with or without amifostine.
* Compare the feasibility and activity of these regimens in these patients.
* Determine the toxicity of paclitaxel and carboplatin in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to WHO performance status (0 vs 1 vs 2), response to induction chemotherapy (complete vs partial vs stable disease vs not evaluable), and participating center.

Patients receive induction chemotherapy comprising paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Patients with a complete or partial response after 2 courses of induction chemotherapy receive 2 additional courses before randomization. Patients with stable disease after 2 courses of induction chemotherapy or who cannot be evaluated after 1 course proceed directly to randomization. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cisplatin IV on days 1, 22, and 43. Patients also undergo radiotherapy daily 5 days a week for 6.5 weeks.
* Arm II:Patients receive amifostine subcutaneously daily. Patients receive chemotherapy and radiotherapy as in arm I.

Patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 41-93 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed undifferentiated nasopharyngeal cancer (UNPC)

  * Locoregionally advanced disease

    * T2b, N1 (greater than 3 cm) or N2
    * T3, N1 (greater than 3 cm) or N2
    * T4, N1 (greater than 3 cm) or N2
    * Any T, N3
  * No squamous cell histology
* At least 1 unidimensionally measurable target lesion

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
* No evidence of distant metastases
* No signs or symptoms of CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 15 to 70

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 150,000/mm^3
* Hemoglobin at least 12 g/dL

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN

Renal:

* Creatinine clearance at least 70 mL/min
* Calcium normal

Cardiovascular:

* No hypotension or hypertension requiring therapy
* No prior myocardial infraction
* No pre-existing uncontrolled cardiac disease
* No signs of cardiac failure
* No rhythm disturbances requiring medication

Other:

* No sensory neuropathy grade 2 or greater unless due to cranial nerve
* No uncontrolled infections
* No sensitivity to aminothiol compounds
* No other malignancy within the past 5 years except adequately controlled carcinoma in situ of the cervix or basal cell or squamous cell skin cancer
* No psychological, familial, sociological, or geographical condition that would preclude study
* Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* No prior chemotherapy for UNPC

Endocrine therapy:

* No concurrent hormonal therapy except corticosteroids for antiemetic prophylaxis

Radiotherapy:

* No prior radiotherapy for UNPC

Surgery:

* No prior surgery for UNPC except cervical lymphadenectomy

Other:

* At least 1 month since prior investigational agent
* No other concurrent anticancer drugs

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2001-07; Primary Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Licitra, MD, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (13):
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- France (2):
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
- Italy (4):
  - Ospedale Santa Croce, Cuneo
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa (Genova)
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Milano (Milan)
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
- Spain (2):
  - Hospital General de Jerez, Jerez de la Frontera
  - Hospital Universitario 12 de Octubre, Madrid
- Istanbul University-Institute of Oncology, Istanbul, Turkey (Türkiye)
- Beatson Oncology Centre, Glasgow, Scotland, United Kingdom